CLINICAL TRIAL: NCT06566586
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQB3702 Tablets Combined With Immunochemotherapy for the Treatment of B-cell Lymphoma
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of TQB3702 Tablets Combined With Immunochemotherapy for the Treatment of B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3702-II-02
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-04

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3702 tablets+Chemotherapy regimen (Experimental): TQB3702 tablets 200mg, every 4 weeks for a treatment cycle.
  Chemotherapy regimen：Every 3 or 4 weeks is a treatment cycle, with 6 or 12 cycles of combination therapy
  Interventions: Drug: TQB3702 tablets+Chemotherapy regimen

INTERVENTIONS:
Drug: TQB3702 tablets+Chemotherapy regimen — TQB3702 tablets: Tyrosine kinase inhibitor；
  Chemotherapy regimen：inhibiting tumor cell proliferation, suppressing DNA synthesis, inducing cell apoptosis, enhancing immune system function, and inhibiting angiogenesis；

SUMMARY:
To evaluate the efficacy and safety of TQB3702 tablets combined with immunochemotherapy for the treatment of B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and the compliance was good;
* Age: 18 years old ≤ age (when signing the informed consent) ≤75 years old; Eastern cooperative oncology group (ECOG) score: 0-2; Expected survival of more than 3 months;
* Histologically confirmed B-cell lymphomas of the following types that meet the 2022 World Health Organization (WHO) diagnostic criteria:

  1. Relapsed/refractory indolent B-cell lymphoma
  2. Diffuse large B cell lymphoma（DLBCL）
* Previous treatment: Relapsed/refractory inert B-cell lymphoma: have received at least one previous line of systemic standard therapy
* Have at least one measurable lesion.
* The main organs function well.
* Female subjects of reproductive age should agree to use contraception (such as Iuds, contraceptives, or condoms) during the study period and for 6 months after the end of the study; Have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Male subjects should agree to use avoidance during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Have had or are currently suffering from other malignant tumors within 3 years prior to the first medication.
* Known or suspected central nervous system (CNS) aggression.
* Relapsed/refractory inert B-cell lymphoma: previous allogeneic hematopoietic stem cell transplantation, or autologous hematopoietic stem cell transplantation within 3 months before the first treatment;
* Recurrent/refractory indolent B-cell lymphoma: toxic reactions that do not return to ≤ National Cancer Institute standard for common toxic reactions (NCI-CTC) AE Grade 1 due to any previous treatment, excluding hair loss and fatigue;
* Have multiple factors that affect oral drug absorption (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
* Received major surgical treatment or significant traumatic injury within 28 days before the start of study treatment;
* Hyperkinetic/venous thrombosis events occurred within 6 months before the first medication;
* Have a history of psychotropic drug abuse and can not quit or have mental disorders;
* Subjects with any severe and/or uncontrolled disease;
* Received live vaccine or messenger ribonucleic acid (mRNA) vaccine within 4 weeks before the first dose, or planned to receive live vaccine or mRNA vaccine during the study;
* Participated in clinical trials of other antitumor drugs within 4 weeks before the first medication;
* Subjects who, in the judgment of the investigator, have concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are not suitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.
Complete response rate (CRR) | Up to 2 years
  The rate of complete tumor remission

SECONDARY OUTCOMES:
Adverse events (AE) and serious adverse events (SAE) | Baseline to up to 28 days
  Incidence and severity of adverse events (AE) and serious adverse events (SAE), as well as abnormal laboratory test indicators
ORR and CRR at the end of combination therapy | Up to 1 year
  Objective response rate and complete remission rate at the end of combination therapy.
Progression-free survival (PFS) | Up to 2 years
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Duration of response (DOR) | Up to 2 years
  The period from the participants first achieving CR or PR to disease progression
Overall survival (OS) | Up to all-cause death
  OS is defined as the time from the first administration to all-cause death
1-year PFS and OS | Up to 1 year
  1-year Progression-free survival and Overall survival rates
2-years PFS and OS | Up to 2 years
  2-years Progression-free survival and Overall survival rates

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Cancer Hospital Chinise Academy of Medical Sciences, Beijing, Beijing Municipality
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guigang City People's Hospital, Guigang, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - PuYang AnYang District Hospital, Anyang, Henan
  - Puyang People's Hospital, Puyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hosiptal, Tongji Medical College, Huazhong University of Science And Technolocy, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital and The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The second Hospital of dalian, Dalian, Liaoning
  - The Second Affiliated Hospital Of Xi'an Jiaotong University(Xibei Hospital), Xi'an, Shaanxi
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang